CLINICAL TRIAL: NCT04697186
Title: Efficacy and Safety of Berberine Hydrochloride, Amoxicillin and Rabeprazole Triple Therapy in the First Eradication of Helicobacter Pylori
Brief Title: Helicobacter Pylori Eradication With Berberine Plus Amoxicillin Triple Therapy Versus Bismuth-containing Quadruple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20202119
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Dyspepsia; Chronic Gastritis; Gastric Cancer; Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Berberine
MeSH Terms: conditions — Dyspepsia; Stomach Neoplasms | interventions — Berberine; Amoxicillin; Rabeprazole; Clarithromycin; Bismuth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine , amoxicillin and rabeprazole triple therapy (Experimental): Berberine 300mg three time daily for 14days, amoxicillin 1000 mg and rabeprazole 10 mg by mouth, twice daily for 14 days.
  Interventions: Drug: Berberine; Drug: Amoxicillin; Drug: Rabeprazole
- Bismuth-containing Quadruple Therapy (Active Comparator): amoxicillin 1000 mg，clarithromy 500mg，rabeprazole 10 mg, and Bismuth 220mg by mouth, twice daily for 14 days.
  Interventions: Drug: Amoxicillin; Drug: Clarithromycin; Drug: Rabeprazole; Drug: Bismuth

INTERVENTIONS:
Drug: Berberine — berberine , amoxicillin and rabeprazole triple therapy group: given for 14 days at a dose of berberine 100 mg 3 tablets TID, amoxicillin 500 mg 2 capsules BID ，rabeprazole 10 mg BID.
  Arms: berberine , amoxicillin and rabeprazole triple therapy
Drug: Amoxicillin — berberine , amoxicillin and rabeprazole triple therapy group: given for 14 days at a dose of berberine 100 mg 3 tablets TID, amoxicillin 500 mg 2 capsules BID ，rabeprazole 10 mg BID.
  Other Names: Amoxy
  Arms: berberine , amoxicillin and rabeprazole triple therapy
Drug: Rabeprazole — berberine , amoxicillin and rabeprazole triple therapy group: given for 14 days at a dose of berberine 100 mg 3 tablets TID, amoxicillin 500 mg 2 capsules BID ，rabeprazole 10 mg BID.
  Other Names: Pariet
  Arms: berberine , amoxicillin and rabeprazole triple therapy
Drug: Amoxicillin — Bismuth-containing Quadruple Therapygroup: given for 14 days at a dose of amoxicillin 500 mg 2 capsules BID ，clarithromycin 500mg BID ,rabeprazole 10 mg BID and bismuth 110 mg 2 capsules BID
  Other Names: Amoxy
  Arms: Bismuth-containing Quadruple Therapy
Drug: Clarithromycin — Bismuth-containing Quadruple Therapygroup: given for 14 days at a dose of amoxicillin 500 mg 2 capsules BID ，clarithromycin 500mg BID ,rabeprazole 10 mg BID and bismuth 110 mg 2 capsules BID
  Other Names: Krashen
  Arms: Bismuth-containing Quadruple Therapy
Drug: Rabeprazole — Bismuth-containing Quadruple Therapygroup: given for 14 days at a dose of amoxicillin 500 mg 2 capsules BID ，clarithromycin 500mg BID ,rabeprazole 10 mg BID and bismuth 110 mg 2 capsules BID
  Other Names: Pariet
  Arms: Bismuth-containing Quadruple Therapy
Drug: Bismuth — Bismuth-containing Quadruple Therapygroup: given for 14 days at a dose of amoxicillin 500 mg 2 capsules BID ，clarithromycin 500mg BID ,rabeprazole 10 mg BID and bismuth 110 mg 2 capsules BID
  Arms: Bismuth-containing Quadruple Therapy

SUMMARY:
This study aims at evaluating efficacy and safety of berberine hydrochloride, amoxicillin and rabeprazole triple therapy versus bismuth-containing quadruple therapy(amoxicillin, clarithromycin, rabeprazole and bismuth) in the first eradication treatment of H. pylori. It is hypothesized that berberinehydrochloride, amoxicillin and rabeprazole triple therapy is non-inferior to bismuth-containing quadruple therapy. Patients diagnosed with H. pylori infection will be randomly divided into one of the above treatments. At week 6 follow-up visits, a urea breath test，rapid urease test or helicobacter pylori stool antigen test will be performed to confirm eradication.

DETAILED DESCRIPTION:
Detailed Description:

The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 14 days and subjects eligibility will be evaluated after signing informed consent. One of urea breath test，rapid urease test or helicobacter pylori stool antigen test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 13 and 17.

Follow-up: includes one visits. Approximately 28 days after the end of treatment. Eradication of H. Pylori will be confirmed by one of urea breath test，rapid urease test or helicobacter pylori stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18~70,both gender.
2. Patients with upper gastrointestinal symptoms and with documented H.pylori infection who did not receive Helicobacter pylori eradication treatment;
3. Patients are willing to receive eradication treatment.
4. Women of childbearing age were required to use medically acceptable contraceptive methods during and 30 days after the trial.

Exclusion Criteria:

1. Patients are excluded if they have previously used antibiotics to eradicate adequately recorded infection with H. pylori.
2. Patients with contraindications or allergies to the study drug.
3. Severe organ damage and complications (such as liver cirrhosis, uremia, etc.), severe or unstable cardiopulmonary or endocrine diseases.
4. Constant use of anti-ulcer drugs ( including taking proton-pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test),antibiotics or bismuth complexes (more than 3 times /1 month before screening).
5. Patients were diagnosed with gastroduodenal ulcer and MALTlymphoma.
6. Pregnant or lactating women.
7. Underwent upper gastrointestinal Surgery.
8. Patients with moderate to severe dysplasia or high degree of intraepithelial neoplasia.
9. Patients have symptom of dysphagia.
10. Evidence of bleeding or iron efficiency anemia.
11. A history of malignancy.
12. Drug or alcohol abuse history in the past 1 year.
13. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs,anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
14. Patients who has psychological problem or poor compliance.
15. Enrolled in other clinical trials in the past 3 months.
16. Refuse to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative urea breath test，rapid urease test or helicobacter pylori stool antigen test 28 days after the end of treatment.

SECONDARY OUTCOMES:
symptoms effective rate | 14 days of treatment, and 28 days after treatment
  Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment.
  Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%.
  Total score = frequency + severity.
  Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence.
  Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3 presenting most severe
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No